CLINICAL TRIAL: NCT04499885
Title: Potential Role of Gastric Lavage by Paraffin Oil in Acute Aluminum Phosphide Poisoning: A Randomized Controlled Clinical Trial
Brief Title: Potential Role of Gastric Lavage by Paraffin Oil in Acute Aluminum Phosphide Poisoning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ghada protocol
Record Dates: First submitted 2020-08-01; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Toxicity, Drug
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Gastric Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paraffin oil gastric lavafe (Active Comparator): Gastric lavage will be initiated with 50 mL of Paraffin oil and 50 mL of sodium bicarbonate solution
  Interventions: Device: Paraffin oil gastric lavage
- Saline gastric lavage (Active Comparator): Gastric lavage with saline and sodium bicarbonate
  Interventions: Device: Gastric lavage with saline and sodium bicarbonate 8.4%

INTERVENTIONS:
Device: Paraffin oil gastric lavage — Gastric lavage will be initiated with 50 mL of Paraffin oil and 50 mL of sodium bicarbonate solution
  Other Names: Paraffin oil
  Arms: Paraffin oil gastric lavafe
Device: Gastric lavage with saline and sodium bicarbonate 8.4% — Gastric lavage with saline and sodium bicarbonate 8.4%
  Other Names: Saline gastric lavage
  Arms: Saline gastric lavage

SUMMARY:
Potential Role of Gastric Lavage by Paraffin Oil in Acute Aluminum Phosphide Poisoning.

DETAILED DESCRIPTION:
The study aims to investigate the Potential Role of Gastric Lavage by Paraffin Oil in Acute Aluminum Phosphide Poisoning: A Randomized Controlled Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* • Patients with symptomatic acute aluminum phosphide poisoning

Exclusion Criteria:

* • Pregnant and lactating women

  * Asymptomatic patients with history of acute aluminum phosphide exposure.
  * Patients with ingestion or exposure to other substances in addition to aluminum phosphide.
  * Patients with other major medical conditions (e.g. cardiovascular disease, renal or hepatic failure).
  * Patients with previous medical intervention (had gastric lavage in any medical center before admission).
  * Patients with disturbed consciousness level
  * Patients with post cardiac arrest cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of deaths | 6 months
  The number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Ezzat Helal, Ass. Prof., Principal Investigator — Forensic medicine Department- Tanta University; Ayman Nagy, ass. Prof., Principal Investigator — Forensic medicine Department- Tanta University; Ghada N. El-Sarnagawy, ass. Prof., Principal Investigator — Forensic medicine Department- Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No